CLINICAL TRIAL: NCT01775033
Title: Regionalized Pediatric Emergency Care in Rural Pennsylvania: the Optimizing Utilization and Rural Emergency Access for Children Study
Brief Title: Regionalized Pediatric Emergency Care in Rural Pennsylvania
Acronym: OUTREACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeremy Kahn, Associate Professor of Critical Care, Medicine and Health Policy & Management, University of Pittsburgh
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H3AMC24076; NCT02306408 (obsolete NCT alias)
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Emergencies
Keywords: Pediatrics; Emergency medical services; Emergency Treatment; Telemedicine
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multicomponent intervention (Experimental): Hospitals in the experimental arm will receive a four-component intervention that integrates local education, community outreach, telemedicine and protocolized triage and transport
  Interventions: Other: Multicomponent intervention
- Control (No Intervention): Hospitals in the control arm will receive usual care.

INTERVENTIONS:
Other: Multicomponent intervention — Develop, implement and evaluate an organized system of regional pediatric emergency care in rural Western Pennsylvania using four pillars: education, community, protocolized triage and transport, and telemedicine.
  Arms: Multicomponent intervention

SUMMARY:
The overall goal of this project is to develop and evaluate an organized, regional system of pediatric emergency care in rural western Pennsylvania.

DETAILED DESCRIPTION:
The OUTREACH project will develop, implement and evaluate an organized system of regional pediatric emergency care in rural western Pennsylvania. Toward that end the investigators have developed three broad goals: (1) to define the key barriers and potential solutions to regionalized pediatric emergency care through community stakeholder engagement; (2) to implement a regionalized system of pediatric emergency care using education, community outreach and telemedicine; and (3) evaluate the impact of the system on health care access and outcomes for rural children. The investigators will implement the intervention in a sample of rural hospitals in Pennsylvania using a staggered roll-out design, and compare outcomes of children seen in these hospitals to similar matched hospitals in the state, using Pennsylvania state Medicaid data to evaluate the impact of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pennsylvania
* Medicaid beneficiary
* Less than or equal to 18 years of age

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5000 (Actual)
Dates: Start 2012-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Average distance from home to the nearest facility with specialized pediatric emergency care capabilities | One-year
  This population-based outcome will act as a measure of access and relates to HRSA Maternal Child Health Bureau performance measure AHS-8 and AHS-9 (access to pre-hospital EMS and wait times)

SECONDARY OUTCOMES:
Incidence of emergency transfers to CHP after an index community ED visit | 90 days
Incidence of emergency transfers to CHP that do not result in a hospital admission | 90 days
Total health care encounters outside the county within three months after an index community ED visit | 90 days
Mortality after an index community ED visit for specified high-risk conditions (trauma, sepsis, and in the chronic disease population) | 90 days
  These outcomes will address our goal to increase child health and related to the HRSA Maternal Child Health Bureau performance measures MICH-1,2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy M Kahn, MD, MS, Study Director — University of Pittsburgh
Locations (1):
- University of Pittburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Lorch SA, Myers S, Carr B. The regionalization of pediatric health care. Pediatrics. 2010 Dec;126(6):1182-90. doi: 10.1542/peds.2010-1119. Epub 2010 Nov 1. PMID 21041285
- [Background] Berger E. Growing pains: Report notes pediatric emergencies need greater emphasis. Ann Emerg Med. 2006 Aug;48(2):143-4. doi: 10.1016/j.annemergmed.2006.06.024. No abstract available. PMID 16953527